CLINICAL TRIAL: NCT01155349
Title: Cognitive Speed of Processing Training Among Persons With Parkinson's Disease
Brief Title: Brain Fitness in Parkinson's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Principal Investigator, Jerri D. Edwards, Associate Professor, University of South Florida
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: USF105832
Record Dates: First submitted 2010-06-29; First posted 2010-07-01 (Estimated); Last update posted 2012-12-10 (Estimated); Status verified 2012-12

CONDITIONS: Parkinson's Disease
Keywords: brain fitness; cognitive training; cognitive intervention; speed of processing training; Parkinson's disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- InSight Brain Fitness (Experimental)
  Interventions: Behavioral: InSight
- No contact-control (Placebo Comparator)
  Interventions: Other: No contact-control group

INTERVENTIONS:
Behavioral: InSight — A cognitive intervention designed to enhance speed of visual processing.
  Arms: InSight Brain Fitness
Other: No contact-control group — No contact-control group.
  Arms: No contact-control

SUMMARY:
The purpose of this study is to examine the feasibility and potential effectiveness of a cognitive training program among persons with Parkinson's disease. It is hypothesized that individuals with PD will be able to complete and benefit from the intervention.

DETAILED DESCRIPTION:
Parkinson's Disease (PD) affects about 1 million individuals in the United States. In addition to the typical motor dysfunction, PD also affects cognition and vision, even in early stages of the disease, impairing instrumental activities of daily living such as driving. Reduced cognitive speed of processing, or bradyphrenia, strongly contributes to cognitive decline in PD. Recent research has demonstrated that interventions can enhance cognitive speed of processing, protect against further cognitive decline, and improve the everyday functioning of relatively healthy, older adults. However, the potential of such training techniques to enhance cognitive functions among subpopulations with different disease states, such as PD, has not been thoroughly investigated. The proposed study will further examine the feasibility and test the efficacy of a well-established cognitive training tool among individuals in the early stages of PD who have not been diagnosed with dementia. A variety of factors have been found to influence cognitive performance among persons with PD and may moderate their ability to benefit from cognitive training such as age at disease onset, disease duration, manifestation, severity, and medication use as well as concomitant depression. These factors along with demographic variables will be evaluated as moderators of training benefit. Baseline cognitive assessments will be completed among seventy-five individuals with PD who will be randomized to cognitive training or a treatment-delayed control condition. The efficacy of training to immediately enhance cognitive functioning will be evaluated through a post-training (or equivalent delay) assessment. Disease and demographic factors that may impact the efficacy of cognitive training for persons with PD will be examined in relation to training gains. Considering that cognitive function among individuals with PD is a strong predictor of everyday functioning and subsequent need for long term care, enhancing cognitive function of individuals with PD through training has great potential to prolong such persons' productivity, independence, and quality of life. The information gained from this study will be useful for identifying individuals with PD who are most likely to benefit from cognitive training as well as the development, refinement, and implementation of appropriate cognitive interventions for this population.

ELIGIBILITY:
Inclusion Criteria:

* Criteria will be age 40 years or older and clinical diagnosis of idiopathic PD in Hoehn and Yahr stages 1 to 3, and on a stable medication regimen (no expected changes in next six months). Subjects with random or severe motor fluctuations and dyskinesias will be excluded. Further inclusion criteria will be no diagnosis of dementia nor evidence of severe dementia that may limit ability to benefit from training, and adequate visual acuity to view testing and training stimuli (far visual acuity >= 20/80).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2009-07; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Useful Field of View | 3 and 6 months
  A measure of visual processing speed independent of motor speed.

SECONDARY OUTCOMES:
Depressive Symptoms | 3 and 6 months
  GDS and CES-D
CSRQ | 3 and 6 months
  Quality of Life measure

CONTACTS AND LOCATIONS:
Overall Officials: Jerri D Edwards, Ph.D., Principal Investigator — University of South Florida
Locations (1):
- University of South Florida, Tampa, Florida, United States